CLINICAL TRIAL: NCT01281605
Title: Comparison of Two Titration Programs of Adding Insulin Detemir to Oral Antidiabetic Drugs in Poorly Controlled Type 2 Diabetes Patients
Brief Title: Comparison of Two Titration Programs of Adding Insulin Detemir to OADs in Poorly Controlled Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sung-Chen Liu, Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10M MHIS112
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Basal insulin; Insulin detemir; Insulin titration algorithm
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active titration algorithm (Active Comparator): titrate insulin dose by contacting with investigator by telephone weekly.
  Interventions: Behavioral: Active titration algorithm
- Usual titration algorithm (Experimental): contact with investigator only at routine study visit.
  Interventions: Behavioral: Usual titration algorithm

INTERVENTIONS:
Behavioral: Active titration algorithm — Patients in active titration algorithm group will contact with investigator by telephone weekly to self-adjust the insulin dose till they achieve the target of FPG(<110mg/dl).
  Other Names: Insulin detemir active titration algorithm
  Arms: Active titration algorithm
Behavioral: Usual titration algorithm — All patients will be instructed to self-measure fasting capillary blood glucose. The dose of insulin detemir will be adjusted based on the average of three consecutive FPG values. the daily insulin dose should be increased by 2 IU/day if the FPG>=110mg/dL, and by 4 IU/day if the FPG>=180 mg/dL without any intervening hypoglycemic episodes; or it should be decreased by 2 or 4 IU/day if the FPG < 70 mg/dL.
  Other Names: Insulin detemir usual titration algorithm
  Arms: Usual titration algorithm

SUMMARY:
This study compared the effectiveness and safety of two treatment algorithms for insulin detemir initiation and titration: active titration algorithm (performed by investigator weekly) versus usual titration algorithm (performed by study subjects weekly) in patients with type 2 diabetes poorly controlled by OADs.

DETAILED DESCRIPTION:
This is a 24-week, prospective, open-label, randomized, parallel-group study conducted in approximately 200 patients with type 2 diabetes in the Taiwan. The effectiveness of insulin detemir will be assessed at baseline and at 12 and 24 weeks after initiation of study prescription. The safety will be followed during the 24-week study period.

Inclusion criteria:

Patients must meet all of the following criteria:

1. Men and women with type 2 diabetes.
2. 20 years of age.
3. Patients who have received stable doses of any OADs for at least 10 weeks prior to the screening visit.
4. Patients with inadequate glycemic control (HbA1C >=7% and < 11%).
5. Patients who are willing and able to cooperate with study and give signed informed consent.

After enrollment, eligible patients will be randomized in a 1:1 ratio to one of the following titration algorithms:

* Active titration algorithm: contact with investigator by telephone weekly.
* Usual titration algorithm: contact with investigator only at routine study visit.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria:

1. Men and women with type 2 diabetes.
2. 20 years of age.
3. Patients who have received stable doses of any OADs for at least 10 weeks prior to the screening visit.
4. Patients with inadequate glycemic control (HbA1C >=7% and < 11%).
5. Patients who are willing and able to cooperate with study and give signed informed consent.

Exclusion Criteria:

1. Patients with type 1 diabetes.
2. Renal dialysis patients.
3. History of hypoglycemia unawareness.
4. Patients who had received any insulin for more than 2 weeks or who have received insulin treatment within 4 weeks prior to screening visit.
5. Patients who have received any investigational products (drug and device) within 4 weeks prior to screening visit.
6. Patients hypersensitive with insulin detemir or its excipients.
7. Patients who are currently pregnant/lactating,or who are preparing for pregnancy or lactation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To compare the change in HbA1c between two study groups at Week 24. | 24 weeks
  compare the change in HbA1c between two study groups after 24 weeks treatment.

SECONDARY OUTCOMES:
To compare the change in HbA1C between two study groups at Week 12. | 12 weeks
  compare the change in HbA1C between two study groups after 12 of treatment.
To compare the proportion of patients achieving HbA1C <7% at Week 24 | 24 weeks
  compare the proportion of patients achieving HbA1C <7% after 24 weeks treatment
To compare the changes in fasting plasma glucose (FPG) at Week 12 and 24. | 24 weeks
  compare the changes in fasting plasma glucose (FPG) after 12 and 24 treatment.
To compare the change in body weight at each visit | 24 weeks
  compare the change in body weight at each visit
To evaluate the incidence of adverse events. | 24 weeks
  evaluate the incidence of adverse events including hypoglycemia and any other adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chen Liu, MD, Study Chair — Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital; Hui-Fang Chang, MD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital Hsinchu branch; Ke-Yan Wu, MD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital Taitung branch
Locations (3):
- Taiwan (3):
  - Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital Hsinchu branch, Hsinchu
  - Mackay Memorial Hospital, Taipei
  - Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital Taitung branch, Taitung